CLINICAL TRIAL: NCT06687031
Title: Cross Cultural Adaptation and Psychometric Properties of Urdu Version of Fall Risk Questionnaire
Status: Not yet recruiting | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR & AHS/24/0231
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Older People
Keywords: Fall risk questionnaire, Psychometric, Reliability, Translation, Validity,

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fall is an event that result a person coming to rest inadvertently on the ground or floor or other lower level. Fall and fall related injuries are very common in older population. Fall can cause potentially life threatening events that can lead to hospitalization and increase cost and burden on society and even lead to the death. Several tools are use for fall risk assessment but in current study we will use fall risk questionnaire that is translated in many languages that is Arabic, Persian, Brazil Turkish and Chinese but no study has translated the fall risk questionnaire into Urdu language. The objective of current study is to translate the fall risk questionnaire into Urdu to determine its reliability and validity in Urdu speaking older population of Pakistan. .

The study will be cross sectional in which original English version of questionnaire will be translated into Urdu language using five steps as described by beaten. The study will be conducted at Service hospital Lahore and Mian Munshi District Head Quarter hospital Lahore. In this study sample size of 120 participants is calculated based on previously published guidelines and according to previously described inclusion and exclusion criteria individuals with age 65 or above 65 who can speak and understand urdu will be included and individuals with any neurological or orthopedic problem that disturb their walking and balance will be excluded. For data collection two physiotherapist (assessor A and assessor B) will examine the enrolled individual separately using fall risk questionnaire, time up and go test, berg balance scale, 5 times sit to stand test and the assessor B will conduct examination 2 hours later to check the inter rater reliability .To determine the intra rater reliability assessor A will again conduct the examination after 7 to 10 days. After collection of data the statistical data analysis will be performed of the collected data using SPSS version 21 with p value will be set to be statistically significant at 0.05 to check the reliability and validity of the Urdu version of fall risk questionnaire. Pearson r will show the co relation of fall risk questionnaire with Berg balance scale, time up and Go test and five times sit to stand test and cronbach's value will show the internal consistency and interclass correlation coefficient ICC will assess the test retest reliability of fall risk questionnaire.

DETAILED DESCRIPTION:
Fall is define as an event which causes a person to unintentionally rest on the ground or floor or lower level. Fall is a movement down that happens due to the gravity. It is the act of going down from upright position suddenly and involuntarily .Fall can occur in every population like in pediatric adults and in geriatric population. But it is very common in older adults aged 65 years and above. The aging population constitute a large and increasing percentage of the world population .When people grow older they experience deterioration in their physiological system and functional status decline until they become frail.

One out of four individual with age 65 years or above experiences at least one fall in every year.(1) In a review of 104 studies with a total sample people of the world is 26.5%(95%CI 23.4-29.8)(2)the present studies show that prevalence of fall in Pakistan is 42.6%(3).In studies 62% of older people were found to have one to two falls resulting in increase risk of fall and consequent injuries. Death in 84.6% of older adult result from fall related injuries than from other causes and 38.19% hospital admission are consequences of fall .

There are different causes of fall it may be due to intrinsic factors( age, impaired balance and gait, decrease muscle strength, impaired vision, cognition, dizziness, depression) and extrinsic factors(medications, opioids, antidepressant, anesthesia ,,inappropriate shoes household setting unsafe furniture, dim light ,presence of loss rug, lack of safety handrails).

Fall can result in fractures, particularly of the hip, wrist, arm, and ankle that can be debilitating and may require surgery or prolonged rehabilitation. It can lead to head injuries, including concussions and traumatic brain injuries (TBIs), which can have serious long-term consequences, especially in older adults. Fall can cause bruises, sprains, strains, and other soft tissue injuries, which may be painful and limit mobility. After experiencing a fall, older adults may develop a fear of falling again,(bisphobia) leading to decreased activity levels, loss of confidence, and social isolation. Severe falls can result in a loss of independence if they lead to disabilities or impairments that affect daily activities and mobility. It often result in hospitalization, which can lead to complications such as infections, pressure ulcers, and deconditioning, particularly in older adults with pre-existing health conditions.. Fall can have psychological effects, including anxiety, depression, and a decrease in overall well-being, affecting both the individual and their caregivers or family members Several tools are commonly use for fall risk assessment in the older population that include downton fall risk, mobility interaction fall chart, St.Thomas risk assessment tool, time up and Go test TUG, Berg balance scale BBS, five times sit to stand test(5TSTST) performance oriented mobility assessment POMA, Fall efficacy scale FES the, Morse Fall scale, Hendrich ll fall risk model, fall risk assessment tool (FRAT) the mini BESTest (Mini balance evaluation system test).(4) In current study we will use fall risk questionnaire FRQ for assessment of the fall in older population. Rubenstein at al developed and validated the simple, brief, and fast 12-question self-rated Fall Risk Questionnaire(FRQ).It has 12 yes or no question the scoring of yes for the first two question is 2 (yes=2)while yes=1 in the remaining 10 questions and No=0 in all 12 questions. If the participants score is 4 or greater than 4 it means he is at risk of fall.

Fall risk questionnaire is translated in to many languages due to its reliability and validity it is translated into Arabic, Thai, brazil, Turkish, Protégées, Persian and Chinese language. More than 65 million people worldwide speak Urdu, mostly from Pakistan and India. Moreover, Urdu is national language of Pakistan. In Pakistan most of the people don't read or understand English very well specially the older population, so different questionnaire should be translated into Urdu. Therefore, the current study is aim at determining the validity and reliability of Urdu translation of fall risk questionnaire FRQ in the context of its acceptability, internal consistency, reliability, interrater reliability, and construct validity in older population.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

* Both male and female gender will be included.
* Age of the individuals will be 65 to 80 year.
* Individuals can ambulate without using assistive devices.
* Individuals can speak Urdu.
* Individuals can understand the command.
* Individuals who don't have communication problem.
* Individuals having mini mental score equal and greater than 24.

Exclusion Criteria:

Individuals with neurological and orthopedic problem that disturb their balance and walking.

* Individuals with cardiovascular problem or uncontrolled hypertension.
* Individual who are alcoholic or any drug addict.
* Individuals who undergo chemotherapy or radiotherapy .

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Study Population: older population
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Urdu version of Fall Risk Questionnaire | 12 weeks
  FRQ is very reliable and valid tool for assessing the risk of fall in older population. It is translated into different languages (Thai, Brazil, Chinese, Persian, Turkish, Arabic) due to its reliability and validity. It has 12 yes or no questions that assess different fall related risk factors in older adults. The answers are scored as yes=2 or no=0 for the first two questions while in remaining ten questions yes=1. Total score of fall risk questionnaire is 14 the score of 4 or greater than 4 indicates that older adult is at risk of falling.
Berg balance scale | 12 weeks
  It is reliable and valid tool to determine the balance of the individual through series of predetermined tasks. There are different version of berg balance scale (Brazilian, Persian, Russian, Itallian, Urdu). It has 14 items list (sit to stand , stand unsupported, sitting unsupported, sitting to stand transfers, standing with eyes closed, standing with feet close together, reaching forward with outstretched arm, retrieving objects from the floor, turning to look behind, turn 360 degree, place alternate foot on the floor, stand on one foot) with each item consists of five points ranging from 0 to 4. 0 means lowest level of function while 4 means highest level of function and it takes about 20 minutes to complete. Equipments require during performance are stop watch, a ruler,2 standard chairs one with arm arrest and one without arm rest a footstool or step and 15 ft walkway. A score of 56 indicates functional balance and a score of <45 indicates individual may be at gr
Time up and Go test | 12 weeks
  Time up and go test is used to determine dynamic balance and it is a a reliable tool for assessing balance in older adult age above 65. In this test participant is sitting on a standard arm chair and we ask the patient to stand up when the instructor say go and then walk to the 3 meter line on the floor at normal pace and then turn and walk back to the chair at the normal pace and sit down again. On the word go start the timer on the stop watch and stop the timer when patient sit back on the chair and record the time. If patient score is equal or greater than 12 then he is at risk of falling.
Five Times Sit to Stand test | 12 weeks
  It is a reliable test to measure the strength of lower limb muscle along balance in older population . It is devised by Causka and McCarty. In this test patient is sitting in standard height chair and his both hands are placed on the opposite shoulder with back straight and instructed to do sit to stand five times as quickly as possible at the count of go and without their back or leg resting on the chair between the interval of repetition. Timer should start when instructor says start and stops when individual's buttock touches the seat of the chair after the last repetition. Inability to complete five repetition without assistance or use of upper extremity support indicates failure of the test any modification should be documented. The normal score for the 60 to 69 years age group is 11.4 sec and 12.6 sec for 70 to 79 years age group and 14.8 sec for 80 to 89 years age group.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif Shaffi, PhD-PT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubenstein LZ, Vivrette R, Harker JO, Stevens JA, Kramer BJ. Validating an evidence-based, self-rated fall risk questionnaire (FRQ) for older adults. J Safety Res. 2011 Dec;42(6):493-9. doi: 10.1016/j.jsr.2011.08.006. Epub 2011 Nov 17. PMID 22152267
- [Background] Kitcharanant N, Vanitcharoenkul E, Unnanuntana A. Validity and reliability of the self-rated fall risk questionnaire in older adults with osteoporosis. BMC Musculoskelet Disord. 2020 Nov 18;21(1):757. doi: 10.1186/s12891-020-03788-z. PMID 33208120
- [Background] Argyrou C, Dionyssiotis Y, Galanos A, Kantaidou I, Vlamis J, Triantafyllopoulos IK, Lyritis GP, Dontas IA, Chronopoulos E. Development and validation of a fall risk Questionnaire in Greek community-dwelling individuals over 60 years old. J Frailty Sarcopenia Falls. 2022 Sep 1;7(3):133-146. doi: 10.22540/JFSF-07-133. eCollection 2022 Sep. PMID 36119553
- [Background] Alharbi AA, Al Amer HS, Albalwi AA, Muthaffar MY, Alshehre YM, Albalawi HF, Alshaikhi TE. Cross-Cultural Adaptation and Psychometric Properties of the Arabic Version of the Fall Risk Questionnaire. Int J Environ Res Public Health. 2023 Apr 21;20(8):5606. doi: 10.3390/ijerph20085606. PMID 37107888
- [Background] Salari N, Darvishi N, Ahmadipanah M, Shohaimi S, Mohammadi M. Global prevalence of falls in the older adults: a comprehensive systematic review and meta-analysis. J Orthop Surg Res. 2022 Jun 28;17(1):334. doi: 10.1186/s13018-022-03222-1. PMID 35765037
- [Background] Ambrose AF, Paul G, Hausdorff JM. Risk factors for falls among older adults: a review of the literature. Maturitas. 2013 May;75(1):51-61. doi: 10.1016/j.maturitas.2013.02.009. Epub 2013 Mar 22. PMID 23523272